CLINICAL TRIAL: NCT01965028
Title: Effectiveness of Daily Bi-temporal Transcranial Random Noise Stimulation in Patients With Chronic Tinnitus
Brief Title: Daily Bi-temporal Transcranial Random Noise Stimulation in Tinnitus
Acronym: tRNS-tin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., M.D., Ph.D., University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Reg-tRNS01
Record Dates: First submitted 2013-10-14; First posted 2013-10-18 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Tinnitus
Keywords: tinnitus; transcranial random noise stimulation; tRNS; auditory cortex; non-invasive brain stimulation
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation

ARMS (1):
- Transcranial random noise stimulation (tRNS) (Experimental): High frequency tRNS (Neuroconn, Eldith DC-Stimulator Plus): 100-650Hz, 2mA, 20min, 10s ramp time, left and right auditory cortex, 5x7cm electrode with the inferior middle part over T3/T4
  Interventions: Device: Transcranial random noise stimulation (tRNS)

INTERVENTIONS:
Device: Transcranial random noise stimulation (tRNS) — High frequency tRNS (Neuroconn, Eldith DC-Stimulator Plus): 100-650Hz, 2mA, 20min, 10s ramp time, left and right auditory cortex, 5x7cm electrode with the inferior middle part over T3/T4 Arms: tRNS

SUMMARY:
Stimulation of the left and right auditory cortex with daily transcranial random noise stimulation (tRNS) is used to modulate the neural pathways involved in chronic tinnitus.

DETAILED DESCRIPTION:
Tinnitus is the phantom auditory perception of sound in the absence of an external or internal acoustic stimulus. It is a frequent problem which can interfere significantly with the ability to lead a normal life. Tinnitus has been shown to be generated in the brain, as a result of functional reorganization of auditory neural pathways and the central auditory system. These changes are represented by hyper-activity and hyper-synchronicity in the auditory pathway. Treatment remains difficult. Non-invasive brain stimulation methods has shown to be effective in the treatment of chronic tinnitus with moderate effect size. Preliminary data presented on international conferences suggest the use of transcranial random noise stimulation (tRNS) over both auditory cortices as new and highly effective treatment. High-frequency (hf; 100-650Hz) tRNS might be highly effective in tackling hyper-synchronised cell assemblies. Daily Hf-tRNS (2 weeks) will be examined with regard to feasibility, safety and clinical efficacy in patients suffering from chronic tinnitus in an one-arm pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bothersome, subjective chronic tinnitus
* Diagnosis: Duration of tinnitus more than 6 months

Exclusion Criteria:

* Objective tinnitus
* Irregular head shap below the electrodes
* Eczema on the head
* Treatable cause of the tinnitus
* Involvement in other treatments for tinnitus at the same time
* Clinically relevant psychiatric comorbidity
* Clinically relevant unstable internal or neurological comorbidity
* History of or evidence of significant brain malformation or neoplasm, head injury
* Cerebral vascular events
* Neurodegenerative disorder affecting the brain or prior brain surgery
* Metal objects in and around body that can not be removed
* Pregnancy
* Alcohol or drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of treatment responders (response: Tinnitus Questionnaire total score reduction ≥ 5, contrast baseline versus end of treatment/week 12) | Week 12

SECONDARY OUTCOMES:
Change of tinnitus severity as measured by the Tinnitus Questionnaire | Week 2
Change of tinnitus severity as measured by the Tinnitus Questionnaire | Week 4
Change of tinnitus severity as measured by the Tinnitus Questionnaire | Week 12
Change of tinnitus severity as measured by the Tinnitus Numeric Rating Scales | Week 2
Change of tinnitus severity as measured by the Tinnitus Numeric Rating Scales | Week 4
Change of tinnitus severity as measured by the Tinnitus Numeric Rating Scales | Week 12
Change of depressive symptoms as measured by the Major Depression Inventory | Week 2
Change of depressive symptoms as measured by the Major Depression Inventory | Week 4
Change of depressive symptoms as measured by the Major Depression Inventory | Week 12
Change in quality of life as measured by the WHOQoL-Bref | Week 2
Change in quality of life as measured by the WHOQoL-Bref | Week 4
Change in quality of life as measured by the WHOQoL-Bref | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, MD, Ph.D., Principal Investigator — University of Regensburg
Locations (1):
- University of Regensburg - Dept of Psychiatry, Regensburg, Germany

REFERENCES:
- [Derived] Kreuzer PM, Poeppl TB, Rupprecht R, Vielsmeier V, Lehner A, Langguth B, Schecklmann M. Daily high-frequency transcranial random noise stimulation of bilateral temporal cortex in chronic tinnitus - a pilot study. Sci Rep. 2019 Aug 22;9(1):12274. doi: 10.1038/s41598-019-48686-0. PMID 31439873